CLINICAL TRIAL: NCT02681380
Title: Impact of a Relation Training, Balint-like, on Empathy of Medical Student in the 4th Year.
Brief Title: Impact of a Relation Training on Empathy of Medical Student
Acronym: EMPATHIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: University Paris 7 - Denis Diderot (Other); University of Paris 13 (Other)
Responsible Party: Principal Investigator, Céline Buffel du vaure, MD, University of Paris 5 - Rene Descartes
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 01004
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Empathy
Keywords: simulated patient; Balint; empathy; medical student
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relation learning (Experimental): Participants of this group will benefit form a specific learning on relation, Balint like. They will have 7 sessions during 3 months.
  Interventions: Other: Relation learning
- Control group (Placebo Comparator): Participants of this group will have no learning related to relation with patient.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Relation learning — Seven session are planned. Each will be supervised by a senior, trained to supervised Balint group.
  Arms: Relation learning
Other: Control group — No session will be planned for the participants.
  Arms: Control group

SUMMARY:
Empathy is an important skill to learn for medical student. However, learning empathy remain difficult. The investigators aim was to assess the efficacy of a specific training, Balint like, on the empathy abilities of medical students in the 4th year. The investigators planned a randomized controlled trial in 3 universities.

ELIGIBILITY:
Inclusion Criteria:

* Medical student in the 4th year

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Care | Two weeks after the last session
  Scale to measure empathy by a simulated patient, during a simulated visit

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jaury, Principal Investigator — University Paris 5

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buffel du Vaure C, Lemogne C, Bunge L, Catu-Pinault A, Hoertel N, Ghasarossian C, Vincens ME, Galam E, Jaury P. Promoting empathy among medical students: A two-site randomized controlled study. J Psychosom Res. 2017 Dec;103:102-107. doi: 10.1016/j.jpsychores.2017.10.008. Epub 2017 Oct 17. PMID 29167035